CLINICAL TRIAL: NCT00070954
Title: Ginkgo Biloba for ECT-induced Memory Deficits
Brief Title: Ginkgo Biloba to Improve Short-Term Memory Losses Associated With Electroconvulsive Therapy (ECT)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: John S. Markowitz, Pharm.D., Medical Univ of SC
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R21AT000939-01A1 (NIH); R21AT000939-01A1 (NIH)
Record Dates: First submitted 2003-10-09; First posted 2003-10-13 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2008-08

CONDITIONS: Memory, Short-Term
Keywords: ECT; Memory; Ginkgo biloba
MeSH Terms: interventions — Ginkgo Extract

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- 2 (Placebo Comparator): look-alike placebo
  Interventions: Other: matched placebo
- Ginkgo Biloba (Active Comparator): Compared to placebo
  Interventions: Drug: ginkgo biloba

INTERVENTIONS:
Drug: ginkgo biloba — EgB 761
  Other Names: ginkgo
  Arms: Ginkgo Biloba
Other: matched placebo — Inactive look-alike placebo
  Arms: 2

SUMMARY:
Electroconvulsive therapy (ECT) is an effective treatment for severe or medication-resistant depression and other psychiatric disorders. A common side effect of ECT is problems with short-term memory during treatment. This study will test whether taking ginkgo biloba (GB) prior to and during the course of ECT will lessen the effects of ECT on short-term memory.

DETAILED DESCRIPTION:
ECT is a safe and effective modern treatment for severe depression and other psychiatric conditions. An estimated 100,000 treatments occur per year in the United States. ECT's most bothersome adverse effect is memory loss, with all patients receiving ECT experiencing some degree of short-term cognitive impairment. At present there are no known effective pharmacologic treatments to prevent or improve ECT-induced cognitive dysfunction. Preliminary research has shown the herbal preparation GB aids cognitive function and memory in both patients with dementia and in normal volunteers. This study will investigate the utility and safety of GB to minimize the cognitive impairment typically associated with ECT.

Participants in this study will be randomly assigned to receive either twice-daily GB or placebo. Participants will begin taking GB or placebo as soon as consent is obtained and baseline testing is completed in order to reach steady-state plasma levels of GB prior to ECT. Patients will undergo cognitive testing at specified intervals following ECT. The final study visit will occur one week after a participant's final ECT treatment.

ELIGIBILITY:
Inclusion Criteria

* DSM-IV diagnosis of major depressive episode, unipolar or bipolar, without psychotic features
* Receiving ECT for depression
* Able to complete detailed neuropsychological testing

Exclusion Criteria

* Psychotic symptoms
* Lifetime history of schizophrenia, schizoaffective disorder, or mental retardation
* Diagnosis of anxiety disorder, obsessive-compulsive disorder, or eating disorder within 1 year of study entry
* Delirium, dementia, or amnestic disorder
* Any active general medical condition or central nervous system disease which could affect cognition or response to treatment
* Diagnosis of active substance abuse or dependence within 6 months of study entry
* ECT within 6 months of study entry
* Known or suspected coagulation disorder
* Anticoagulation or antiplatelet medications, including warfarin, aspirin, clopidogrel, and ticlopidine
* Thiazide diuretics, selective serotonin reuptake inhibitors, trazodone, antipsychotic medications, herbal medications, or other nutritional supplements
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2003-02; Primary Completion 2005-01 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Modified Mini-Mental State Examination | 2009
Rey Auditory Verbal Learning Test | 2009
Autobiographical Memory Inventory | 2003-2009
Spitzer Uniscale of Quality of Life(Uni) | 2--3-2009
Health Status Questionnaire | 2003-2009

CONTACTS AND LOCATIONS:
Overall Officials: John S. Markowitz, PharmD, Principal Investigator — Medical University of South Carolina; Charles H. Kellner, M.D., Principal Investigator — UMDNJ - NJ Medical School; Thomas W Uhde, MD, Study Chair — Medical University of South Carolina
Locations (1):
- UMDNJ - NJ Medical School, Newark, New Jersey, United States